CLINICAL TRIAL: NCT04461366
Title: Monopolar Radiofrequency Versus Pulsed Dye Laser for Treatment of Acne Scars: A Randomized Clinical Trial
Brief Title: Monopolar Radiofrequency Versus Pulsed Dye Laser for Treatment of Acne Scars
Acronym: MRFPDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002410
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Acne Atrophica
Keywords: Acne scars; Monopolar radiofrequency; Pulsed dye laser
MeSH Terms: interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monopolar radiofrequency (MRF) group (Experimental): Monopolar Radiofrequency Diathermy (LVT-250, Korea) was used at average energy160-180 W, main power 50/60 Hz, 40˚C ~ 45˚C Temperature, RF output 470 kHz, 20 mm electrode size.
  Interventions: Device: Monopolar radiofrequency
- Pulsed dye laser (PDL) group (Active Comparator): Flash lamp pulsed dye laser; Candela SPTL-1 (Candela Corp., Wayland, Mass.) with the following parameters: (585nm wavelength, 450 msec pulse duration, 6.5 to 7.5 J/cm² energy density and 5or 7mm spot size).
  Interventions: Device: Pulsed dye laser

INTERVENTIONS:
Device: Monopolar radiofrequency — The RF electrode was moved randomly for 30 seconds over each scar. The total duration of the treatment session is only 5 minutes for each cheek. It takes 15 minutes if the forehead and 2 cheeks are affected.
  Arms: monopolar radiofrequency (MRF) group
Device: Pulsed dye laser — PDL was applied for the affected areas with no pre-treatment regimens or topical anaesthetics. There was no requirement for skin cooling.
  Arms: Pulsed dye laser (PDL) group

SUMMARY:
Background: The acne scar is a common disorder characterized by skin eruption or abnormalities on face, chest, and/or back in the adolescence which affect the cosmetic appearance.

Purpose: The main aim of this study was to investigate whether monopolar radiofrequency (MRF) or pulsed dye laser (PDL) is more effective in the cases suffering from acne scars in the form of reducing acne scars and improving the cosmetic appearance.

DETAILED DESCRIPTION:
Thirty patients suffering from moderate or severe acne scars were randomly assigned into two equal groups. Group A (MRF group): received 2 sessions per week with MRF for 8 weeks. Group B (PDL group): received 1 session per week with PDL for 8 weeks. The severity of acne scars was assessed before and after treatment by using the clinical evaluation scale for acne scarring (ECCA) scale and the self-assessment of clinical acne-related scars (SCARS) scale. Quality of life and the emotional impact of acne scars were evaluated by the facial acne scar quality of life (FASQoL) scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to severe acne scar
* Patients with acne scar in the face

Exclusion Criteria:

* Smokers and alcohol drinker
* Patients who had a history of diabetes, circulatory or sensory disorders
* Patients who had a history of frequent sunburns
* Patients with nodulocystic acne

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — adolescents
Enrollment: 30 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
acne scars severity by investigator | after 8 weeks of intervention
  Clinical evaluation scale for acne scarring. Using this scale, the type of scar was defined by the qualitative descriptions of scars, which is then accompanied by a numerical score (0-4) and then multiplied by (15-50) which is a weighting factor of clinical severity, the total possible score is from 0 to 540. Higher score means worse outcome while lower score means better out come.
acne scars severity by the participant | after 8 weeks of intervention
  Self-assessment of clinical acne-related scars questionnaire. It consists of 5-items with 1 hypothesized domain which asks patients to assess acne scars severity as seen in the mirror. The total possible score is from 0- 20. Higher score means worse outcome while lower score means better out come.

SECONDARY OUTCOMES:
emotional, social functioning and work/school effect of scars | after 8 weeks of intervention
  Facial acne scar quality of life scale. It is a tool formed of 10-items with 3 domains to assess the emotional, social functioning and work/school effect of scars on a 5-point rating scale The total possible score is from 0- 40. Higher score means worse outcome while lower score means better out come.

CONTACTS AND LOCATIONS:
Overall Officials: Nesma M Allam, PhD, Principal Investigator — lecturer at faculty of physical therapy
Locations (1):
- Radwa T Elshorbagy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
I will share data 6 months after publication
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: study protocol